CLINICAL TRIAL: NCT05211453
Title: A Randomised Comparison of Left and Right Sided Approaches to Ablation of the Atrioventricular Junction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Sussex Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Rick Veasey, Principal Investigator, East Sussex Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S001
Record Dates: First submitted 2021-11-09; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrioventricular node
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right sided atrioventricular node ablation (Active Comparator): Right sided atrioventricular node ablation
  Interventions: Procedure: atrioventricular node ablation
- Left sided atrioventricular node ablation (Active Comparator): Left sided atrioventricular node ablation
  Interventions: Procedure: atrioventricular node ablation

INTERVENTIONS:
Procedure: atrioventricular node ablation — atrioventricular node ablation

SUMMARY:
This study will compare right sided atrioventricular node ablation to left sided atrioventricular node ablation

DETAILED DESCRIPTION:
Right-sided atrioventricular node ablation has been the initial conventional approach however up to 18.5% of patients require switching to a left sided approach or have a challenging procedure. Previous studies have found that left sided ablation is more efficacious than right-sided ablation requiring less than 5 applications of radiofrequency energy to induce atrioventricular block.

This study will compare right sided atrioventricular node ablation to left sided atrioventricular node ablation

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Referred for atrioventricular node ablation for any such indication

Exclusion Criteria:

* Stroke or transient ischaemic attack (TIA) within 6 months
* Myocardial infarction within 6 months
* Medical conditions limiting expected survival to <1 year
* Moderate to severe aortic stenosis
* History of aortic or mitral valve replacement
* Pregnancy or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of total ablation time required to induce complete atrioventricular node block | intraoperative
  Time in seconds

SECONDARY OUTCOMES:
Comparison of number of RF applications required to induce complete atrioventricular node block | intraoperative
  Comparison of number of RF applications required to induce complete atrioventricular node block
Comparison of total procedure time between the two groups | intraoperative
  Comparison of total procedure time between the two groups
Comparison of radiation exposure between the two groups | intraoperative
  Comparison of radiation exposure between the two groups
Comparison of rate of the escape rhythm after ablation in beats/min | intraoperative
  Comparison of rate of the escape rhythm after ablation in beats/min
Comparison of number of patients requiring crossover to each side | intraoperative
  Comparison of number of patients requiring crossover to each side
Comparison of adverse events / complications between each group | intraoperative
  Comparison of adverse events / complications between each group
Comparison of patient comfort of procedure | intraoperative
  Comparison of patient comfort of procedure using visual analogue scale ( 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Veasey, Principal Investigator — East Sussex Healthcare NHS
Locations (1):
- Eastbourne District General Hospital, Eastbourne, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No